CLINICAL TRIAL: NCT04647799
Title: Electrophysiological Studies Of Induced Forward Head Position And Hand Use Of Mobile Phone
Brief Title: Effect of Use Smartphone in Forward Head Position and Neutral Position on Upper Limbs Nerves
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Karim Samy Ibrahim, principal investigator, MTI University
Other Study IDs: 012/002542
Record Dates: First submitted 2020-09-14; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Mobile Phone Use
MeSH Terms: conditions — Cell Phone Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- forward head position: nerve conduction velocity and f-wave applied to median , ulnar and radial nerve before and after 10,20 and 30 minutes in forward head position while Children will sit on chair with their feet on the ground without any tension, the upper limbs are rested in a table then, the angle between the line passing horizontally from the spinous process of C7 and the line passing between the tragus and spinous process of C7 will be measured by goniometer and goniometer pro application to evaluate the craniovertebral angle recording, we will fix the craniovertebral angle between 40.7° and 43.2°(severe FHP )
  Interventions: Device: smartphone
- neutral position: nerve conduction velocity and f-wave applied to median , ulnar and radial nerve before and after 10,20 and 30 minutes while Children will sit on chair with their feet on the ground with head in anatomical position, the upper are rested in a table and used both hand on touch screen of mobile phone
  Interventions: Device: smartphone

INTERVENTIONS:
Device: smartphone — Samsung A 71
  Other Names: mobile phone

SUMMARY:
To compare between two different positions (forward head position and neutral position) when using mobile phone by hand using nerve conduction velocity and F-wave of upper limb nerves ( ulnar, median and radial) in 4 different times.

DETAILED DESCRIPTION:
PURPOSE:

* To compare between forward head position and hand use of mobile phone on conduction velocity of upper limb nerves
* To investigate the F responses of upper limbs nerves.
* To investigate the compound muscle action potential (CMAP) amplitudes of median nerves

BACKGROUND:

Forward head position may affect the cervical nerve root so it can also affect nerve conduction velocity due to continues stretch on nerves, also the over use of smart phone by hand may be affected the hand nerves, so this study determine which one of them has more influence than the other.

If the forward head position has the worst effect on the upper limb nerves investigators must avoid the incorrect position of the head to avoid stretch and compression of the nerves.

HYPOTHESES:

There are no statistical difference between forward head position and hand use of mobile phone on conduction velocity of the nerves of upper limb.

SUBJECTS:

Normal one hundred fifty non-athketic adolescents of both genders will participate in this study. Their age ranges from 14-18 years.

METHODS FOR ASSESSMENT

1. Electromyography (EMG) will be used to measure nerve conduction velocity, F-wave, motor action potential
2. Soft collar will used to fixed the craniovertebral angle during used mobile phone Universal goniometer
3. Goniometer pro iPhone application

ELIGIBILITY:
Inclusion Criteria:

1. Their ages range from 14-18 years.
2. Not rolled on any regular athletic activity

Exclusion Criteria:

1. Individual with neck pain
2. Congenital deformity for upper limb
3. Peripheral neuropathy due to diabetes mellitus type I
4. Rheumatoid arthritis
5. History of surgical intervention at nerves of the upper extremity

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: normal subjects
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
motor and sensory nerve conduction velocity and f-wave in neutral position | 1 day
  motor and sensory nerve conduction velocity and f-wave will measured to nerves of upper extremities ( median, ulnar and radial nerves) in neutral position by using electrodiagnosis when using mobile phone

SECONDARY OUTCOMES:
motor and sensory nerve conduction velocity and f-wave measured in forward head position during use mobile phone | 1 day
  motor and sensory nerve conduction velocity and f-wave will measured to nerves of upper extremities ( median, ulnar and radial nerves) in forward head position by using electrodiagnosis when using mobile phone

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pysical Therapy, 6 Oct University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT04647799/Prot_ICF_000.pdf